CLINICAL TRIAL: NCT06564623
Title: A Pilot Study of Targeting Driver Oncogenes With a Peptide Vaccine Plus Durvalumab and Tremelimumab for Patients With Biliary Tract Cancers
Brief Title: Targeting Driver Oncogenes With a Peptide Vaccine Plus Durvalumab and Tremelimumab for Patients With Biliary Tract Cancers (BTC)
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: AstraZeneca (Industry); Private Philanthropic Funds (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: J2477; IRB00416341 (Other: Johns Hopkins Medical Institution)
Record Dates: First submitted 2024-08-19; First posted 2024-08-21 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-12

CONDITIONS: Biliary Tract Cancers
Keywords: Biliary Tract Cancer; Duvalumab; Tremelimumab; Immunotherapy; mBTCvax (peptide vaccine + Poly-ICLC (Hiltonol)); Anti PD-L1; Anti-Cytotoxic T-lymphocyte antigen 4 (CTLA-4); Hiltonol; Carcinoma
MeSH Terms: conditions — Biliary Tract Neoplasms; Diabetes Mellitus, Insulin-Dependent, 12; Carcinoma | interventions — Peptides; poly ICLC; durvalumab; tremelimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Arm A - mBTCvax, Durvalumab and Tremelimumab (Experimental)
  Interventions: Drug: mBTC vax [0.3 - 2.4 mg peptide + 0.5 mg Poly-ICLC (Hiltonol)]; Drug: Durvalumab; Drug: Tremelimumab

INTERVENTIONS:
Drug: mBTC vax [0.3 - 2.4 mg peptide + 0.5 mg Poly-ICLC (Hiltonol)] — Patients will receive treatment on Day 1, 8, 15 and 22 of cycle 1 and on day 1 of remaining cycles (C2-C4) in Prime Phase. In the Boost Phase - every 2 cycles (8 weeks) beginning from C6D1.
  Other Names: Peptide + Poly-ICLC (Hiltonol)
Drug: Durvalumab — Patients will receive treatment on Day 1 of each cycle. Durvalumab (1500 mg) will be administered IV every 4 weeks in both the Prime and Boost Phase.
  Other Names: IMFINZI®
Drug: Tremelimumab — Patients will receive treatment on C1D1. Tremelimumab (300 mg) will be administered IV as a single dose on Day 1 of Cycle 1.
  Other Names: IMJUDO®

SUMMARY:
The purpose of this study is to evaluate the safety and the immune response of personalized mutant peptide vaccine with poly-ICLC adjuvant (mBTCvax) in combination with durvalumab and tremelimumab following front-line treatment in patients with advanced stage BTC.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Must have a histologically- or cytologically, proven biliary tract cancer (BTC) previously treated with gemcitabine/cisplatin/anti-PD(L)1 therapy.
* Must have evidence of radiological disease, must accept to have a tumor biopsy of an accessible lesion at baseline and on treatment.
* Must have sufficient archival tumor tissue for next-generation sequencing (NGS) and immune-phenotyping.
* Have a BTC containing at least one of the oncogenic mutation/alterations targeted by the vaccine.
* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1.
* Must have body weight of >30 kg.
* Patients must have adequate organ and marrow function defined by study-specified laboratory tests.
* Patients with chronic or acute hepatitis B virus (HBV) or hepatitis C virus (HCV) infection must have disease controlled prior to enrollment.
* Women of childbearing potential (WOCBP) must have a negative urine or serum pregnancy test.
* For both Women and Men, must use acceptable form of birth control while on study.
* Must have a life expectancy of at least 12 weeks.
* Ability to understand and willingness to sign a written informed consent document.

Exclusion Criteria:

* Participation in another clinical study with an investigational product during the last 2 weeks.
* Patient is expected to require any other form of systemic or localized antineoplastic therapy while on study.
* Any of the following procedures or medications within 2 weeks prior to initiation of study treatment:

  * Systemic or topical steroids at immunosuppressive doses (> 10 mg/day of prednisone or equivalent). The following are exceptions to this criterion:
  * Intranasal, inhaled, topical steroids, or local steroid injections (e.g., intra articular injection)
  * Systemic corticosteroids at physiologic doses not to exceed 10 mg/day of prednisone or its equivalent
  * Steroids as premedication for hypersensitivity reactions (e.g., CT scan premedication)
  * Palliative or adjuvant radiation or gamma knife radiosurgery.
  * Chemotherapy or checkpoint inhibitor targeting anti-Pd1/PD-L1.
* Within 4 weeks prior to initiation of study treatment:

  * Any investigational cytotoxic drug.
  * Any investigational device.
  * Non-oncology vaccines containing live virus.
  * Allergen hyposensitization therapy.
  * Growth factors, e.g. granulocyte-colony stimulating factor (G-CSF), granulocyte macrophage-colony stimulating factor (GM-CSF), erythropoietin.
  * Major surgery.
* Any unresolved toxicity NCI CTCAE Grade ≥2 from previous anticancer therapy with the exception of alopecia, vitiligo, and the laboratory values defined in the inclusion criteria.
* Patients with Grade ≥2 neuropathy will be evaluated on a case-by-case basis after consultation with the Study Physician.
* All AEs while receiving prior immunotherapy must have completely resolved or resolved to baseline prior to screening for this study.
* Must not have experienced a ≥Grade 3 immune related AE or an immune related neurologic or ocular AE of any grade while receiving prior immunotherapy.
* Patients with a history of prior treatment with anti-PD-1 and anti-PD-L1.
* History of severe hypersensitivity reaction to any monoclonal antibodies or related compounds or to any of its components.
* History of leptomeningeal carcinomatosis.
* Patient has a known history or evidence of brain metastases.
* Has an active known or suspected autoimmune disease or which has required systemic therapy in the last 5 years.
* Known history of interstitial lung disease or of (non-infectious) pneumonitis that required steroids or current pneumonitis.
* Has a pulse oximetry < 92% on room air.
* Requires the use of home oxygen.
* Has a known history of Human Immunodeficiency Virus (HIV)/AIDS
* Has active co-infection with HBV (hepatitis B virus) and HCV (hepatitis C virus) or coinfected with HBV and hepatitis delta virus (HDV)
* Uncontrolled intercurrent illness including, but not limited to, uncontrolled infection, symptomatic congestive heart failure, unstable angina, cardiac arrhythmia, metastatic cancer, or psychiatric illness/social situations that would limit compliance with study requirements.
* Patients who have been diagnosed with another cancer or myeloproliferative disorder in the past 5 years requiring systemic therapy or expected to require active therapy within the clinical study period.
* Has a diagnosis of immunodeficiency.
* Presence of any tissue or organ allograft, regardless of need for immunosuppression, including corneal allograft. Patients with a history of allogeneic hematopoietic stem cell transplant will be excluded.
* Any other sound medical, psychiatric, and/or social reason as determined by the Investigator.
* Patient is at the time of signing informed consent a regular user (including "recreational use") of any illicit drugs or had a recent history (within the last year) of substance abuse (including alcohol).
* Patient is unwilling or unable to follow the study schedule for any reason.
* Pregnant or breastfeeding.
* WOCBP and men with female partners (WOCBP) who are not willing to use contraception.
* Evidence of clinical ascites requiring paracentesis in the last 4 weeks.
* History of malignant bowel obstruction.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2025-05-27 (Actual); Primary Completion 2029-05 (Estimated); Study Completion 2029-05 (Estimated)

PRIMARY OUTCOMES:
Number of participants experiencing grade 3 or above drug-related toxicities | 20 Months
  When calculating the incidence of Adverse Events (AE), each AE (as defined by NCI CTCAE v5.0) will be counted only once for a given subject.
Maximum percentage change in interferon-producing mutant-specific cluster of differentiation 8 (CD8) and cluster of differentiation 4 (CD4) T cells. | Baseline to 20 weeks post vaccination (baseline, 20 weeks)
  Evaluated by the maximal percent change in interferon-producing mutant-specific CD8 and CD4 T cells within 20 weeks post-vaccination compared to pre-vaccination baseline.

SECONDARY OUTCOMES:
Progression Free Survival (PFS) | 4 years
  PFS is defined as the number of months from the date of first vaccine dose until the date of disease progression using RECIST 1.1 criteria or death due to any cause, whichever occurs first, for BTC patients. PFS will be censored at the date of the last scan for subjects without documentation of disease progression at the time of analysis. Per RECIST 1.1 criteria, Complete Response (CR) = disappearance of all target lesions, Partial Response (PR) is =>30percent decrease in sum of diameters of target lesions, Progressive Disease (PD) is >20percent increase in sum of diameters of target lesions, Stable Disease (SD) is <30percent decrease or <20percent increase in sum of diameters of target lesions. Estimation based on the Kaplan-Meier curve.
Overall Survival (OS) | 4 years
  OS will be defined as the number of months from the date of first vaccine dose until date of death due to any cause. OS will be censored on the date the subject was last known to be alive for subjects without documentation of death at time of analysis. Estimation based on the Kaplan-Meier curve.

CONTACTS AND LOCATIONS:
Overall Officials: Marina Baretti, MD, Principal Investigator — SKCCC Johns Hopkins Medical Institution
Locations (1):
- SKCCC Johns Hopkins Medical Institution, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No